CLINICAL TRIAL: NCT03289962
Title: A Phase 1a/1b Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of RO7198457 as a Single Agent and in Combination With Atezolizumab in Patients With Locally Advanced or Metastatic Tumors
Brief Title: A Study of Autogene Cevumeran (RO7198457) as a Single Agent and in Combination With Atezolizumab in Participants With Locally Advanced or Metastatic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO39733; 2017-001475-23 (EudraCT Number)
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Melanoma; Non-Small Cell Lung Cancer; Bladder Cancer; Colorectal Cancer; Triple Negative Breast Cancer; Renal Cancer; Head and Neck Cancer; Other Solid Cancers
Keywords: Neoantigen; Personalized; Atezolizumab; Immunotherapy; Anti-PDL1; Checkpoint Inhibitor
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Kidney Neoplasms; Head and Neck Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1a Flat Dose Escalation: Autogene Cevumeran (Experimental): Participants will receive autogene cevumeran at escalated dosages.
  Interventions: Drug: Autogene cevumeran
- Phase 1b Flat Dose Escalation: Autogene Cevumeran + Atezolizumab (Experimental): Participants will receive autogene cevumeran at escalated dosages along with atezolizumab at a fixed dose of 1200 milligrams (mg)
  Interventions: Drug: Autogene cevumeran; Drug: Atezolizumab
- Phase Ib: Dose Exploration: Autogene Cevumeran + Atezolizumab (Experimental): Non-small cell lung cancer (NSCLC) or melanoma cancer immunotherapy (CIT)-treated participants will receive autogene cevumeran (at dosage lower than maximum tolerated dose [MTD] based on available safety data) along with atezolizumab at a fixed dose of 1200 mg.
  Interventions: Drug: Autogene cevumeran; Drug: Atezolizumab
- Phase 1b Expansion: Autogene Cevumeran + Atezolizumab (Experimental): Participants with different indications as per inclusion criteria will receive autogene cevumeran (at multiple dose levels below MTD based on available safety data) along with atezolizumab at a fixed dose of 1200 mg.
  Interventions: Drug: Autogene cevumeran; Drug: Atezolizumab
- Phase 1b Expansion: Autogene Cevumeran + Atezolizumab (Serial Biopsy) (Experimental): CIT-naive patients with selected tumor types who consent to optional serial biopsies will receive autogene cevumeran (at multiple dose levels below MTD based on available safety data) along with atezolizumab at a dixed dose of 1200 mg.
  Interventions: Drug: Autogene cevumeran; Drug: Atezolizumab

INTERVENTIONS:
Drug: Autogene cevumeran — Autogene cevumeran will be administered by intravenous (IV) infusion, in 21-day cycles.
  Other Names: RO7198457
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion on Day 1 of every 21-day cycle.
  Other Names: Tecentriq; RO5541267; MPDL3280A; An engineered anti-PDL1 antibody
  Arms: Phase 1b Expansion: Autogene Cevumeran + Atezolizumab; Phase 1b Expansion: Autogene Cevumeran + Atezolizumab (Serial Biopsy); Phase 1b Flat Dose Escalation: Autogene Cevumeran + Atezolizumab; Phase Ib: Dose Exploration: Autogene Cevumeran + Atezolizumab

SUMMARY:
This is a Phase 1a/1b, open-label, multicenter, global, dose-escalation study designed to evaluate the safety, tolerability, immune response, and pharmacokinetics of autogene cevumeran (RO7198457) as a single agent and in combination with atezolizumab (MPDL3280A, an engineered anti-programmed death-ligand 1 [anti-PD-L1] antibody).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>=12 weeks)
* Adequate hematologic and end-organ function
* Measured or calculated creatinine clearance >=50 milliliters per minute (mL/min) on the basis of the Cockcroft-Gault glomerular filtration rate estimation

Cancer-Specific Inclusion Criteria:

* Participants with histologic documentation of locally advanced, recurrent, or metastatic incurable malignancy that has progressed after at least one available standard therapy; or for whom standard therapy has proven to be ineffective or intolerable, or is considered inappropriate; or for whom a clinical trial of an investigational agent is a recognized standard of care
* Participants with confirmed availability of representative tumor specimens in formalin-fixed, paraffin-embedded (FFPE) blocks (preferred), or sectioned tissue
* Participants with measurable disease per RECIST v1.1

Additional Inclusion Criteria for Participants in Each Indication-Specific Exploration/Expansion Cohort of Phase 1b:

* NSCLC Cohorts (CIT-Naive): Participants with histologically confirmed incurable, advanced NSCLC not previously treated with anti-PD-L1/PD-1 and/or with anti-CTLA-4 (investigational or approved), for whom a clinical trial of an investigational agent in combination with an anti-PD-L1/PD-1 antibody is considered an acceptable treatment option (if CIT [including anti-PD-L1/PD-1 agents] is approved as treatment for NSCLC by local regulatory authorities).
* NSCLC Cohort (CIT-Treated): Participants with histologically confirmed incurable, advanced NSCLC previously treated with anti-PD-L1/PD-1 with or without anti-CTLA-4 (investigational or approved)
* Triple negative breast cancer (TNBC) Cohort (CIT-Naive): Participants with histologically confirmed incurable, advanced estrogen receptor (ER)-negative, progesterone receptor-negative, and human epidermal growth factor receptor 2 (HER2)-negative adenocarcinoma of the breast (triple-negative) not previously treated with anti-PD-L1/PD-1 and/or anti-CTLA-4 (investigational or approved)
* Colorectal cancer (CRC) Cohort (CIT-Naive): Participants with histologically confirmed incurable, advanced adenocarcinoma of the colon or rectum not previously treated with anti-PD-L1/PD-1 and/or anti-CTLA-4 (investigational or approved)
* Head and neck squamous cell carcinoma (HNSCC) Cohort (CIT-Naive): Participants with histologically confirmed inoperable, locally advanced or metastatic, recurrent, or persistent HNSCC (oral cavity, oropharynx, hypopharnyx, or larynx) not amenable to curative therapy not previously treated with anti-PD-L1/PD-1 and/or anti-CTLA-4 (investigational or approved)
* Urothelial carcinoma (UC) Cohort (CIT-Naive): Participants with histologically confirmed incurable, advanced transitional cell carcinoma of the urothelium including renal pelvis, ureters, urinary bladder, and urethra, not previously treated with anti-PD-L1/PD-1 with or without anti-CTLA-4 (investigational or approved), for whom a clinical trial of an investigational agent in combination with an anti-PD-L1 antibody is considered an acceptable treatment option, if CIT (including anti-PD-L1/PD-1 agents) is approved as treatment for UC by local regulatory authorities
* UC Cohort (CIT-Treated): Participants with histologically confirmed incurable advanced transitional cell carcinoma of the urothelium (including renal pelvis, ureters, urinary bladder, and urethra) previously treated with anti-PD-L1/PD-1 with or without anti-CTLA-4 (investigational or approved)
* Renal cell carcinoma (RCC) Cohort (CIT-Naive): Participants with histologically confirmed incurable, advanced RCC with component of clear cell histology and/or component of sarcomatoid histology not previously treated with anti-PD-L1/PD-1 and/or anti-CTLA-4 (investigational or approved)
* Melanoma Cohort (CIT-Naive in metastatic setting): Participants with histologically confirmed incurable, advanced melanoma not previously treated with anti-PD-L1/PD-1 and/or anti-CTLA-4 (investigational or approved) in the metastatic setting
* Melanoma Cohort (CIT-Treated): Participants with histologically confirmed incurable, advanced melanoma previously treated with anti-PD-L1/ or PD-1 with or without CTLA-4 (investigational or approved)

Additional Inclusion Criteria for Participants in the Serial-Biopsy Expansion Cohort of Phase 1b:

* Participants must have one of the locally advanced or metastatic solid tumor types specified in the protocol.
* Participants must have accessible lesion(s) that permit a total of two to three biopsies (pretreatment and on-treatment) or one biopsy (on-treatment, if archival tissue can be submitted in place of a pre-treatment biopsy) without unacceptable risk of a significant procedural complication. RECIST lesions should not be biopsied.

Exclusion Criteria:

* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, and inherited liver disease or current alcohol abuse
* Major surgical procedure within 28 days prior to Cycle 1, Day 1, or anticipation of need for a major surgical procedure during the course of the study
* Any other diseases, metabolic dysfunction, physical examination finding, and/or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or may render the participant at high risk from treatment complications
* Previous splenectomy
* Known primary immunodeficiencies, either cellular (e.g., DiGeorge syndrome, T-negative severe combined immunodeficiency [SCID]) or combined T- and B-cell immunodeficiencies (e.g., T- and B-negative SCID, Wiskott Aldrich syndrome, ataxia telangiectasia, common variable immunodeficiency)
* Any medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study Cancer-Specific Exclusion Criteria
* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, and/or radiotherapy, within 3 weeks prior to initiation of study treatment, with the exceptions as mentioned in the protocol
* Eligibility based on prior treatment with CIT depends on the mechanistic class of the drug and the cohort for which the participant is being considered, as described below. In addition, all criteria pertaining to adverse events attributed to prior cancer therapies must be met

All Cohorts (Dose-Escalation in Phase 1a and Dose-Escalation, Backfill, and Expansion in Phase 1b):

* Prior neoantigen-specific or whole-tumor cancer vaccines are not allowed, with the exception as specified in protocol
* Prior treatment with cytokines is allowed provided that at least 6 weeks or 5 half-lives of the drug, whichever is shorter, have elapsed between the last dose and the proposed Cycle 1, Day 1
* Prior treatment with immune checkpoint inhibitors, immunomodulatory monoclonal antibody (mAbs), and/or mAb-derived therapies is allowed provided that at least 6 weeks (Phase 1a) or 3 weeks (Phase 1b) have elapsed between the last dose and the proposed Cycle 1, Day 1, with the exceptions as specified in protocol Phase Ib Dose-Exploration/Expansion Group Only Cohorts
* In the non-melanoma CIT-Naive expansion cohort in Phase Ib, prior treatment with anti-PD-L1/PD-1 and/or anti-CTLA-4 (investigational or approved), is not allowed.
* In the melanoma CIT-naive in metastatic setting expansion cohort in Phase Ib, prior treatment with anti-PD- L1/PD-1 and/or anti-CTLA-4 (investigational or approved) is not allowed. Prior anti-PD-L1/PD-1 and/or anti-CTLA-4 therapy in the adjuvant setting is allowed provided that there is at least a 6-month treatment-free interval between completion of adjuvant therapy and Cycle 1, Day 1.
* Prior treatment with immunomodulators, including toll-like receptor (TLR) agonists, inhibitors of indoleamine 2,3-dioxygenase (IDO)/ tryptophan-2,3-dioxygenase (TDO), or agonists of OX40, is allowed provided that at least 5 half-lives of the drug or a minimum of 3 weeks have elapsed between the last dose of the prior treatment and the proposed Cycle 1, Day 1, with the exception as specified in protocol
* Any history of an immune-mediated Grade 4 adverse event attributed to prior CIT (other than endocrinopathy managed with replacement therapy or asymptomatic elevation of serum amylase or lipase)
* Any history of an immune-mediated Grade 3 adverse event attributed to prior CIT (other than hypothyroidism managed with replacement therapy) that resulted in permanent discontinuation of the prior immunotherapeutic agent and/or occurred less than or equal to (<=) 6 months prior to Cycle 1 Day 1
* Adverse events from prior anti-cancer therapy that have not resolved to Grade <=1 except for alopecia, vitiligo, or endocrinopathy managed with replacement therapy
* All immune-mediated adverse events related to prior CIT (other than endocrinopathy managed with replacement therapy or stable vitiligo) must have resolved completely to baseline
* Primary central nervous system (CNS) malignancy, untreated CNS metastases, or active CNS metastases (progressing or requiring corticosteroids for symptomatic control)
* Leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Malignancies other than disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death
* Uncontrolled hypercalcemia
* Participant has spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >=2 weeks prior to screening

Treatment-Specific Exclusion Criteria:

* History of autoimmune disease with caveats as specified in protocol
* Treatment with monoamine oxidase inhibitors (MAOIs) within 3 weeks prior to Cycle 1, Day 1
* Treatment with systemic immunosuppressive medications within 2 weeks prior to Cycle 1, Day 1
* History of idiopathic pulmonary fibrosis, pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Positive test for human immunodeficiency virus (HIV) infection
* Active hepatitis B, hepatitis C
* Known active or latent tuberculosis infection
* Severe infections within 4 weeks prior to Cycle 1, Day 1
* Recent infections not meeting the criteria for severe infections within 2 weeks prior to Cycle 1, Day 1
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study
* Known hypersensitivity to the active substance or to any of the excipients in the vaccine
* Phase 1b and crossover only: History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins; Known hypersensitivity to Chinese Hamster Ovary (CHO)-cell products; Allergy or hypersensitivity to components of the atezolizumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Phase 1a: Days 1 to 14 / Phase 1b: Days 1 to 21
MTD/Recommended Phase 2 Dose (RP2D) of Autogene Cevumeran | Phase 1a: Days 1 to 14 / Phase 1b: Days 1 to 21
Percentage of Participants with Adverse Events (AEs) | Baseline up to end of the study (up to approximately 3 years)
Percentage of Participants with Immune-Mediated Adverse Events (imAEs) | Baseline up to end of the study (up to approximately 3 years)
Percentage of Participants by Number of Treatment Cycles Received | Baseline up to end of the study (up to approximately 3 years)
Dose Intensity of Autogene Cevumeran | Baseline up to end of the study (up to approximately 3 years)
Change from Baseline in Targeted Vital Signs | Baseline up to end of study (up to approximately 3 years)
Change from Baseline in Targeted Clinical Laboratory Test Results | Baseline up to end of study (up to approximately 3 years)
Change from Baseline in ECGs | Baseline up to end of study (up to approximately 3 years)

SECONDARY OUTCOMES:
Percentage of Participants with Objective Response of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria for Solid Tumors Version 1.1 (RECIST v1.1) | Baseline until 90 days after last dose or initiation of another systemic anti-cancer therapy, whichever occurs first (up to approximately 3 years)
Duration of Response (DoR) According to RECIST v1.1 | From first occurrence of a documented objective response (CR or PR) until disease progression or death due to any cause, whichever occurs first (up to approximately 3 years)
Percentage of Participants with Objective Response of CR or PR According to Immune-Modified RECIST | Baseline until 90 days after last dose or initiation of another systemic anti-cancer therapy, whichever occurs first (up to approximately 3 years)
DoR According to Immune-Modified RECIST | From first occurrence of a documented objective response (CR or PR) until disease progression or death due to any cause, whichever occurs first (up to approximately 3 years)
Progression-Free Survival (PFS) According to RECIST v1.1 | Baseline until 90 days after last dose or initiation of another systemic anti-cancer therapy, whichever occurs first (up to approximately 3 years)
Overall Survival (OS) | Baseline until 90 days after last dose or initiation of another systemic anti-cancer therapy, whichever occurs first (up to approximately 3 years)
Percentage of Participants with Anti-Drug Antibodies (ADAs) to Atezolizumab | Pre-infusion (0 hr) until 2 months post treatment discontinuation (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (14):
  - HonorHealth Research Institute ? Bisgrove, Scottsdale, Arizona
  - UCSF Comprehensive Cancer Ctr, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University Cancer Center, Smilow Cancer Hospital, New Haven, Connecticut
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Oncology and Hematology Care Eastside, Portland, Oregon
  - Sarah Cannon Res Inst, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (2):
  - UZ Gent, Ghent
  - CHU de Liège (Sart Tilman), Liège
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- Fachklinik für Lungenerkrankungen, Immenhausen, Germany
- Netherlands (2):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (2):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
- Akademiska sjukhuset, Onkologkliniken, Uppsala, Sweden
- United Kingdom (2):
  - Barts & London School of Med, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez J, Powles T, Braiteh F, Siu LL, LoRusso P, Friedman CF, Balmanoukian AS, Gordon M, Yachnin J, Rottey S, Karydis I, Fisher GA, Schmidt M, Schuler M, Sullivan RJ, Burris HA, Galvao V, Henick BS, Dirix L, Jaeger D, Ott PA, Wong KM, Jerusalem G, Schiza A, Fong L, Steeghs N, Leidner RS, Rittmeyer A, Laurie SA, Gort E, Aljumaily R, Melero I, Sabado RL, Rhee I, Mancuso MR, Muller L, Fine GD, Yadav M, Kim L, Leveque VJP, Robert A, Darwish M, Qi T, Zhu J, Zhang J, Twomey P, Rao GK, Low DW, Petry C, Lo AA, Schartner JM, Delamarre L, Mellman I, Lower M, Muller F, Derhovanessian E, Cortini A, Manning L, Maurus D, Brachtendorf S, Lorks V, Omokoko T, Godehardt E, Becker D, Hawner C, Wallrapp C, Albrecht C, Kroner C, Tadmor AD, Diekmann J, Vormehr M, Jork A, Paruzynski A, Lang M, Blake J, Hennig O, Kuhn AN, Sahin U, Tureci O, Camidge DR. Autogene cevumeran with or without atezolizumab in advanced solid tumors: a phase 1 trial. Nat Med. 2025 Jan;31(1):152-164. doi: 10.1038/s41591-024-03334-7. Epub 2025 Jan 6. PMID 39762422